CLINICAL TRIAL: NCT06205745
Title: Quality of Life in Amputated Patients Based on Social Deprivation Factors
Status: Withdrawn | Type: Observational
Why Stopped: Staffing constraints
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202301896
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Amputations for Management of Sarcoma,Trauma,or Chronic Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the quality of life in patients who previously underwent major amputation, and to determine any correlation with social deprivation factors. We hypothesize that patients with increased social deprivation (public or no insurance, lower education, lower income, etc.) will have lower quality of life following amputation.

DETAILED DESCRIPTION:
Amputation remains an important treatment option for patients with sarcoma. While limb salvage procedures have become more widely utilized after the advent of chemotherapy, some patients still require amputation in the management of their disease. Studies have shown that patients with social deprivation factors are at higher risk of presenting with advanced disease, and thus are at increased risk of requiring definitive amputation1-3. Additional research shows amputations are more common in lower socioeconomic status patients4. Whether these procedures are done for trauma or infection, they can have morbid outcomes. Prior literature demonstrates that long-term healthcare costs after amputation are higher than in limb salvage5,6. In some patients, the costs associated with prosthetics may be prohibitive and thus impact quality of life. While many factors are thought to ultimately impact life after amputation7, it remains unclear how social deprivation affects outcomes in patients who undergo an amputation.

Data Collection: Under an approved HIPAA waiver, dependent and independent variables will be collected and retrospectively from a chart review. After we receive the initial request, we will perform a chart review to ensure inclusion/exclusion criteria was met. The following information will be obtained through a combination of the report request and subsequent chart review:

* Demographic Information: Name, MRN, Age, Gender, Insurance Status (private v Medicaid v Medicare v uninsured), Address (including Zip Code), Sarcoma Diagnosis, Amputation Level and Date, Medical Comorbidities
* Survey Information: Current work status and Occupation, Race, Education Level (Highest level degree obtained), Use of prosthesis (and why not if answer is No), Prosthesis Information if yes (Manufacturer and Model), SF-36 Questionnaire, MSTS Tumor Score Questionnaire, Prosthesis Evaluation Questionnaire-Mobility Section (PEQ-MS)

In addition to chart review, subjects will also complete a series of questionnaires to assess outcomes related to surgery. The questionnaires include SF-36 Questionnaire, MSTS Tumor Score Questionnaire, and Prosthesis Evaluation Questionnaire-Mobility Section (PEQ-MS). Prior to contact, subjects will receive a letter (waiver of documentation of informed consent) from the attending physicians describing the study and asking them if they would like to participate in the study by completing the questionnaires and allowing the use of their data for the study. The letter from the attending physicians will also explain that subjects will receive an email or telephone call from a research team member. Subjects will have the opportunity to complete the questionnaire via phone, regular mail, or email using the survey function in RedCap.

Subjects that are willing to complete the questionnaire will be enrolled under a waiver of documentation of informed consent. Subjects that are not willing to complete the questionnaire but will allow their data to be used will be enrolled under a waiver of documentation of informed consent (i.e.: Subject states on the phone they don't want to complete questionnaire, but they give permission for us to retrospectively use their data). Those subjects that have inadequate data or cannot be reached after a reasonable effort will be enrolled under a full waiver of informed consent to use their retrospective data. If subjects indicate on the phone or via email, they do not want their retrospective data used we will withdraw the subject and delete all retrospective data.

Data Analysis: We will perform descriptive statistics on the cohort of patients, as well as report their outcomes. Data will be presented as means and SD for continuous variables and frequencies and percentages for nominal data. We will compare the group of patients with poor outcomes with their counterparts using Student t-tests for continuous variables and Chi square or Fisher exact tests for nominal data.

This study involves minimal risk to patients; however, the patient may experience some psychological and emotional distress when answering questions on the survey. Patients may decline to answer the question or withdraw participation at any time. The investigators will reassure each participant that all survey answers are based on what the participant is feeling and that there is no "correct" answer.

Patients' confidentiality also must be considered during the survey if completed over the phone. However, the study team will establish safeguards to ensure the security and privacy of participants study records. Once all subject data is collected, subject PHI will be removed, and the data will be maintained by using assigned research identification numbers that uniquely identifies each individual. Only IRB approved research personnel will have access to identifiable research data. All recorded data will be labeled using a subject-specific code. A document linking the subject specific code to the name, MRN, relevant dates, e-mail, and telephone number of the subject will be stored securely in a locked cabinet within OSMI and/or electronically on a password-protected server in the University of Florida. All experimental data (defined as all data other than the subject's name, MRN, relevant dates, e-mail address, and telephone number) will only contain the subject-specific code. All data shared with individuals outside the study team will be de-identified, including removal of the subject-specific code

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent major amputation via orthopaedic oncology attending at UF (transtibial, transfemoral, hip disarticulation, transhumeral, or trans-forearm)
* Must be at least 6 months post amputation at the time of survey administration
* Patients undergoing amputation for sarcoma, trauma, or chronic infection

Exclusion Criteria:

* Pediatric patients (<18 years of age)
* Adult patients with the following amputations: ray resection, transmetacarpal, wrist disarticulation, any other amputation distal to the carpi, Syme (ankle disarticulation), Chopart amputation, transmetatarsal, any other amputation distal to the tibia
* Patients undergoing amputations for diabetes or vascular disease
* Patients within 6 months post-operatively from their amputation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 250 patients, 18-90+ years of age, who underwent major amputations for definitive management of their sarcoma, trauma, or chronic infection by our Orthopaedic oncologists (Parker Gibbs Jr., MD, Mark Scarborough, MD, Andre Spiguel, MD). We will determine our participant population using EPIC records of our physicians' case logs. Patients must be at least 6 months postoperative from their amputation to be eligible for contact.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | One visit at least 6 months removed from the amputation
  A survey set of generic, coherent, and easily administered quality-of-life measures.
MSTS Tumor Score Questionnaire | One visit at least 6 months removed from the amputation
  A physician/patient-completed questionnaire designed to assess functional outcome for patients with sarcomas in the extremities.
Prosthesis Evaluation Questionnaire-Mobility Section (PEQ-MS) | One visit at least 6 months removed from the amputation
  A questionnaire that evaluates the perceived potential for mobility using prosthetic devices over the past 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andre Spiguel, MD, Principal Investigator — University of Florida
Locations (1):
- UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided